CLINICAL TRIAL: NCT04176250
Title: A Phase 2a, Dose Escalation, Controlled, Randomized Study to Evaluate Safety, Early Bactericidal Activity (EBA) and Pharmacokinetics of TBA-7371 in Adult Patients With Rifampicin-sensitive Pulmonary Tuberculosis
Brief Title: Early Bactericidal Activity of TBA-7371 in Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gates Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Gates MRI-TBD03-201
Record Dates: First submitted 2019-10-29; First posted 2019-11-25 (Actual); Results first posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Tuberculosis
Keywords: Rifampicin-sensitive pulmonary tuberculosis; TBA-7371; Pulmonary tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- TBA-7371 100 mg QD (Experimental)
  Interventions: Drug: TBA-7371
- TBA-7371 100 mg BID (Experimental)
  Interventions: Drug: TBA-7371
- TBA-7371 200 mg QD (Experimental)
  Interventions: Drug: TBA-7371
- TBA-7371 100 mg TID (Experimental)
  Interventions: Drug: TBA-7371
- TBA-7371 400 mg QD (Experimental)
  Interventions: Drug: TBA-7371
- HRZE (Active Comparator)
  Interventions: Drug: HRZE

INTERVENTIONS:
Drug: TBA-7371 — Participants will receive TBA-7371 oral suspension 100 milligram (mg) once daily (QD) for 14 days.
  Arms: TBA-7371 100 mg QD
Drug: TBA-7371 — Participants will receive TBA-7371 oral suspension 100 mg twice daily (BID) for 14 days.
  Arms: TBA-7371 100 mg BID
Drug: TBA-7371 — Participants will receive TBA-7371 oral suspension 200 mg QD for 14 days.
  Arms: TBA-7371 200 mg QD
Drug: TBA-7371 — Participants will receive TBA-7371 oral suspension 100 mg three times daily (TID) for 14 days.
  Arms: TBA-7371 100 mg TID
Drug: TBA-7371 — Participants will receive TBA-7371 oral suspension 400 mg QD for 14 days.
  Arms: TBA-7371 400 mg QD
Drug: HRZE — Participants will receive Isoniazid [H] / rifampicin [R] / pyrazinamide [Z] / ethambutol [E] (HRZE), a fixed dose combination tablet QD for 14 days, based on weight as 40-54 kilograms (kg): 3 tablets; 55-70 kg: 4 tablets and 71 kg and over: 5 tablets.
  Other Names: Rifafour® e-275
  Arms: HRZE

SUMMARY:
The purpose of this study is to assess the safety, early bactericidal activity (EBA) and pharmacokinetics of TBA-7371 in adult participants with rifampicin-sensitive tuberculosis and select dose regimen(s) for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18 to 60 years of age inclusive at the time of signing the informed consent.
* Body weight within 40 and 100 kilogram (inclusive).
* Untreated, rifampicin-sensitive pulmonary tuberculosis, as defined by all of the following:

  1. isoniazid urine screen negativity
  2. sputum smear positivity on direct microscopy for acid-fast bacilli, defined as at least 1+ on the International Unit Against Tuberculosis and Lung Disease/ World Health Organization scale
  3. chest X-rays which in the opinion of the investigator is consistent with tuberculosis (TB).
  4. Mycobacterium tuberculosis (Mtb) positivity on molecular test (GeneXpert®)
  5. rifampicin sensitivity on molecular test (GeneXpert®).
* Participants must be able to produce at least 10 milliliter of sputum during the overnight sputum collection (day -7 to -3 or day -2 of the Screening Phase).
* Female and male participants should be of non-childbearing potential or using an effective method of birth control.

  * Non-childbearing potential is defined as follows:

    1. participant is not heterosexually active or practices sexual abstinence, OR
    2. female participant or sexual partner has undergone bilateral oophorectomy, bilateral tubal ligation and/or hysterectomy, OR
    3. female participant or sexual partner has been postmenopausal with a history of no menses for at least 12 consecutive months, OR
    4. male participant or sexual partner has undergone vasectomy or bilateral orchidectomy at least three months prior to screening, OR
    5. male participant with pregnant sexual partner (for duration of the study) who does not have any other sexual partners.
  * An effective method of birth control is defined as follows:

    1. double barrier method, which can include any 2 of the following: a male condom, diaphragm, cervical cap, or female condom (male and female condoms should not be used together), OR
    2. barrier method (one of the above) combined with hormone-based contraceptives or an intra-uterine device for the female participant or partner, AND
    3. participant willing to continue practicing one of the above-mentioned birth control methods throughout 14-day Study Treatment Phase and for 4 weeks after the last dose of study medication or discontinuation from study medication in case of early withdrawal.
* Participants must be capable of giving signed informed consent, which includes agreeing to compliance with the requirements and restrictions listed in the informed consent form and the protocol.

Exclusion Criteria:

* Need for immediate effective anti-TB treatment as judged by the investigator.
* Evidence and/or history of extra-thoracic TB (e.g. miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis, ocular TB), as judged by the investigator.
* Evidence and/or history in the last 5 years of one or any combination of the following:

  1. uveitis;
  2. color vision deficiency;
  3. amblyopia;
  4. visual acuity worse than 20/25 after correction in either eye;
  5. any known eye disease or prior eye surgery;
  6. any systemic condition with ocular manifestations (i.e. Marfan, syphilis, diabetes, Beçhet, Vogt-Koyanagi-Harada, Lyme, or chronic inflammatory condition such as sarcoidosis, rheumatoid arthritis, psoriatic arthritis)
* Evidence and/or history in the last 5 years of clinically significant medical condition(s) as judged by the investigator, including malignancies and unstable or uncontrolled hypertension.
* Any current medical, psychiatric, occupational, or substance abuse problems that, in the opinion of the investigator, will make it unlikely that the participant will comply with the protocol.
* For Human Immunodeficiency Virus infected participants:

  1. CD4+ count <350 cells/microliter, OR
  2. Acquired Immune Deficiency Syndrome-defining opportunistic infection or malignancies (except pulmonary TB).
* Seated systolic/diastolic blood pressure assessed as vital sign [i.e. not from electrocardiogram (ECG)] is less than 95/40 millimeters of Mercury (mmHg) or greater than 145/95 mmHg at screening. Out-of-range blood pressure may be repeated twice with at least 5 minutes intervening.
* Seated heart rate assessed as vital sign (i.e. not from ECG) is lower than 40 beats per minute (bpm) or higher than 110 bpm at screening. Out-of-range heart rate may be repeated twice with at least 5 minutes intervening.
* A clinically significant ECG abnormality at screening. NOTE: The following can be considered not clinically significant:

  1. mild first-degree atrio-ventricular block (P-R interval <0.23 seconds);
  2. right or left axis deviation;
  3. incomplete right bundle branch block;
  4. isolated left anterior fascicular block (left anterior hemiblock) in young athletic participants.
* A list of commonly used prohibited medications with the features described below are prohibited:

  * Use of medications active against Mtb within 3 months prior to the first dose of study drug.
  * Use of systemic immunosuppressive medications within 14 days prior to the first dose of study drug.
  * Use of strong inhibitors or strong inducers of cytochrome P450 (CYP) enzymes within 14 days prior to the first dose of study drug.
  * Use of inhibitors of phosphodiesterase (PDE) enzymes within 14 days prior to the first dose of study drug.
  * Use of medications known to affect the eye within 3 months prior to the first dose of study drug.
  * For Human Immunodeficiency Virus positive participants, use of medications listed in the protocol within 3 months prior to the first dose of study drug.
* Participation in other clinical study(-ies) with investigational agent(s) within 6 months prior to trial start.
* The following laboratory values from blood collected during the Screening Phase, which represent Grade 2 or higher abnormalities per Division of Acquired Immune Deficiency Syndrome (DAIDS) Toxicity Table Version 2.1, will be cause for exclusion:

  * Aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase ≥ 2.5x upper limit of normal (ULN) for local laboratory values
  * Total bilirubin ≥ 1.6x ULN
  * Creatinine ≥ 1.3x ULN
  * Hemoglobin < 10 grams per deciliter (g/dL) [male] or 9.5 g/dL [female]
  * White Blood Cells < 2,000 /cubic millimeter (mm3)
  * Platelets ≤ 100,000 /mm3
  * International normalized ratio of prothrombin time (INR) ≥ 1.5x ULN
  * Partial thromboplastin time (PTT) ≥ 1.66 ULN
  * Prothrombin time (PT) ≥ 1.25x ULN
* Grade 2 or higher abnormalities in other laboratory parameters from blood or urine Grade 1 abnormalities, or abnormalities from laboratory parameters not included in the DAIDS Toxicity Table Version 2.1, may lead to exclusion if the investigator considers them clinically significant.
* History of allergy or hypersensitivity to any of the study drugs or related substances.
* Positive urine drug screening for cocaine AND/OR amphetamines AND/OR opiates AND/OR methamphetamines. Note: screening will also be conducted for cannabinoids and results documented in the case report form; however, a positive test for cannabinoids is not an exclusion criterion.
* Female participants currently pregnant or lactating/nursing; OR having positive serum pregnancy test during the Screening Phase OR planning a pregnancy within the 1 month after first dose of study drug.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gates MRI, Study Director — Gates Medical Research Institute
Locations (4):
- South Africa (4):
  - TASK, Bellville, Cape Town
  - University of Cape Town (UCT) Lung Institute, Mowbray, Cape Town
  - The Aurum Institute, Pretoria, Gauteng
  - Perinatal HIV Research Unit (PHRU), Jouberton, North West

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in South Africa.
Pre-assignment Details: This was a dose escalation, controlled, randomized study to evaluate safety, early bactericidal activity (EBA) and pharmacokinetics (PK) of TBA-7371 in adult participants with rifampicin-sensitive pulmonary tuberculosis (TB). Participants were randomized 5:1 to TBA-7371 or HRZE. Data are presented by intervention.
Groups:
- TBA-7371 100 Milligrams (mg) Once Daily (QD): Participants were randomized to receive TBA-7371 oral suspension 100 mg QD for 14 days
- TBA-7371 100 mg Twice Daily (BID): Participants were randomized to receive TBA-7371 oral suspension 100 mg BID for 14 days
- TBA-7371 200 mg QD: Participants were randomized to receive TBA-7371 oral suspension 200 mg QD for 14 days.
- TBA-7371 100 mg Three Times a Day (TID): Participants were randomized to receive TBA-7371 oral suspension 100 mg TID for 14 days.
- TBA-7371 400 mg QD: Participants were randomized to receive TBA-7371 oral suspension 400 mg QD for 14 days.
- Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE): Participants were randomized to receive HRZE, a fixed dose combination tablet QD for 14 days, based on weight as 40-54 kilograms (kg): 3 tablets; 55-70 kg: 4 tablets and 71 kg and over: 5 tablets.
Period: Overall Study
Arm/Group | TBA-7371 100 Milligrams (mg) Once Daily (QD) | TBA-7371 100 mg Twice Daily (BID) | TBA-7371 200 mg QD | TBA-7371 100 mg Three Times a Day (TID) | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Started | 15 | 15 | 15 | 17 | 16 | 15
Completed | 15 | 14 | 14 | 15 | 15 | 13
Not Completed | 0 | 1 | 1 | 2 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Positive CoronaVIrus Disease(COVID)/Severe Acute Respiratory Syndrome CoronaVirus 2(SARS-CoV-2) test | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Randomized in error | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Modified intention-to-treat (mITT) population: included all participants randomly assigned to study intervention, who received at least one dose of the study intervention.
Groups:
- TBA-7371 100 mg QD: Participants were randomized to receive TBA-7371 oral suspension 100 mg QD for 14 days
- TBA-7371 100 mg BID: Participants were randomized to receive TBA-7371 oral suspension 100 mg BID for 14 days
- TBA-7371 100 mg TID: Participants were randomized to receive TBA-7371 oral suspension 100 mg TID for 14 days.
- Total: Total of all reporting groups
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE) | Total
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15 | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.5 (5.10) | 36.3 (10.49) | 27.4 (6.99) | 33.4 (9.27) | 31.3 (12.00) | 27.3 (9.37) | 30.2 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 4 | 6 | 4 | 4 | 25
  Male | 10 | 13 | 11 | 11 | 11 | 11 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 9 | 12 | 9 | 10 | 7 | 9 | 56
  South African Colored | 3 | 2 | 1 | 0 | 2 | 1 | 9
  Mixed Race | 3 | 1 | 5 | 7 | 6 | 5 | 27

OUTCOME MEASURES:

1. Primary Outcome: Average Change Per Day (Slope) of Log Colony Forming Units (CFU) Counts From Day 0 to Day 14 (BACFU [0-14]) to Assess Bactericidal Activity
Description: Overnight sputum samples were collected daily. Bacterial burden was assessed on each sputum sample by CFU on solid culture media. Baseline log10CFU measure was taken as the average of Day -2 and Day -1 log10CFU values. Log10CFU values from subsequent overnight sputum samples (Day 1 to Day 14) were used to assess changes in bacterial burden during the Study Treatment Phase (bactericidal activity). BACFU was the average change in log10CFU count per day over the 14 day Study Treatment Phase. Negative mean BACFU (0-14) values were indicative of a reduction in log10CFU from Baseline, i.e., bactericidal activity. The lower the mean BACFU (0-14) the greater the reduction given it is negative. Positive mean BACFU (0-14) values indicated an increase in log10CFU from Baseline.
Time Frame: Day 0 to Day 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (90% Confidence Interval); unit: log10 CFU per milliliter (/mL) per day
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 15
log10 CFU per milliliter (/mL) per day | -0.039 [-0.074 to -0.005] | -0.086 [-0.123 to -0.049] | -0.065 [-0.101 to -0.029] | -0.130 [-0.163 to -0.098] | -0.096 [-0.130 to -0.061] | -0.203 [-0.238 to -0.168]

2. Primary Outcome: Number of Participants Reporting ≥Grade 3 Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Clinical signs and symptoms that constitute AEs/SAEs were classified by the investigator as mild (Grade 1), moderate (Grade 2), severe (Grade 3), potentially life threatening (Grade 4), death (Grade 5). Number of participants reporting one or more severe AEs (≥grade 3) and SAEs is presented.
Time Frame: Up to Day 15
Population: Safety Population: included all participants randomly assigned to study intervention and who received at least one dose of the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants
  ≥Grade 3 AEs | 0 | 1 | 1 | 2 | 0 | 3
  SAEs | 0 | 1 | 1 | 0 | 0 | 0

3. Secondary Outcome: Average Change Per Day (Slope) of Log CFU Counts From Day 0 to Day 2 (BACFU [0-2]) and From Day 2 to Day 14 (BACFU [2-14]) to Assess Bactericidal Activity
Description: Overnight sputum samples were collected daily. Bacterial burden was assessed on each sputum sample by CFU on solid culture media. Baseline log10CFU measure was taken as the average of Day -2 and Day -1 log10CFU values. Log10CFU values from subsequent overnight sputum samples (Day 1 to Day 14) were used to assess changes in bacterial burden during the Study Treatment Phase (bactericidal activity). BACFU was the average change in log10CFU count per day over the 14 day Study Treatment Phase. Negative mean BACFU (0-2) and BACFU (2-14) values were indicative of a reduction in log10CFU from Baseline, i.e., bactericidal activity. The lower the mean BACFU (0-2) and BACFU (2-14), the greater the reduction given it is negative. Positive mean BACFU (0-2) and BACFU (2-14) values indicated an increase in log10CFU from Baseline.
Time Frame: Day 0 to Day 2 and Day 2 to Day 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (90% Confidence Interval); unit: log10 CFU/mL/day
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 15
log10 CFU/mL/day
  BACFU (0-2) | 0.094 [-0.080 to 0.267] | -0.111 [-0.297 to 0.074] | -0.310 [-0.489 to -0.131] | -0.229 [-0.392 to -0.066] | -0.305 [-0.478 to -0.133] | -0.396 [-0.569 to -0.224]
  BACFU (2-14) | -0.061 [-0.111 to -0.010] | -0.068 [-0.122 to -0.014] | -0.026 [-0.078 to 0.026] | -0.127 [-0.174 to -0.080] | -0.081 [-0.131 to -0.031] | -0.179 [-0.229 to -0.128]

4. Secondary Outcome: Average Change Per Day(Slope)of Time to Sputum Culture Positivity(TTP) in Mycobacteria Growth Indicator Tube (MGIT) System From Day0 to Day14 (BATTP[0-14]),From Day0 to Day2(BATTP[0-2]), and From Day2 to Day14(BATTP [2-14]) to Assess Bactericidal Activity
Description: Overnight sputum samples were collected daily. Bacterial burden was assessed on each sputum sample by time to positivity (TTP; hours) in MGIT system. Baseline TTP measure was taken as the average of Day -2 and Day -1 TTP values. TTP values from subsequent overnight sputum samples (Day 1 to 14) were used to assess changes in bacterial burden during the Study Treatment Phase (bactericidal activity). BATTP was the average change of time to (sputum culture) Positivity (hours) per day in MGIT system per day over 14 days. Positive mean BATTP values were indicative of an increase in TTP from Baseline. The higher the Mean BATTP, the greater the increase given it is positive. Negative mean BATTP values indicated a reduction in TTP from Baseline.
Time Frame: Day 0 to Day 14, Day 0 to Day 2 and Day 2 to Day 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (90% Confidence Interval); unit: Hours per day
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 13 | 15 | 16 | 15 | 15
Hours per day
  BATTP (0-14) | 2.334 [0.533 to 4.135] | 4.143 [2.194 to 6.092] | 3.250 [1.428 to 5.072] | 5.547 [3.803 to 7.291] | 3.767 [1.967 to 5.566] | 13.877 [12.073 to 15.681]
  BATTP (0-2) | 0.961 [-4.214 to 6.135] | 0.902 [-4.697 to 6.502] | 2.749 [-2.485 to 7.982] | 8.633 [3.623 to 13.643] | 12.930 [7.760 to 18.100] | 30.872 [25.690 to 36.054]
  BATTP (2-14) | 2.182 [0.333 to 4.031] | 4.249 [2.247 to 6.250] | 3.811 [1.941 to 5.681] | 5.624 [3.834 to 7.414] | 2.604 [0.757 to 4.452] | 10.660 [8.808 to 12.512]

5. Secondary Outcome: Average Change Per Day (Slope) of the log10 Sputum Lipoarabinomannan (LAM) Measurements From Day 0 to Day 14 (BALAM [0-14]), From Day 0 to Day 2 (BALAM [0-2]) and From Day 2 to Day 14 (BALAM [2-14]) to Assess Bactericidal Activity
Description: Overnight sputum samples were collected daily. Bacterial burden was assessed on each sputum sample by LAM assay in picograms/mL. Baseline log10LAM measure was taken as the average of Day -2 and Day -1 log10LAM values. Log10LAM values from subsequent overnight sputum samples (Day 1 to 14) were used to assess changes in bacterial burden during the Study Treatment Phase (bactericidal activity). Negative mean BALAM values were indicative of a reduction in log10 LAM from Baseline. The lower the Mean BALAM, the greater the reduction given it is negative. Positive mean BALAM values indicated an increase in log10 LAM from Baseline.
Time Frame: Day 0 to Day 14, Day 0 to Day 2 and Day 2 to Day 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (90% Confidence Interval); unit: Picograms per milliliter (pg/mL) per day
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 13 | 15 | 17 | 15 | 15
Picograms per milliliter (pg/mL) per day
  BALAM (0-14) | -0.082 [-0.109 to -0.056] | -0.096 [-0.124 to -0.067] | -0.090 [-0.117 to -0.063] | -0.114 [-0.139 to -0.089] | -0.095 [-0.121 to -0.068] | -0.099 [-0.126 to -0.073]
  BALAM (0-2) | -0.145 [-0.249 to -0.040] | -0.148 [-0.261 to -0.036] | -0.007 [-0.114 to 0.099] | -0.123 [-0.221 to -0.025] | -0.092 [-0.196 to 0.012] | -0.314 [-0.419 to -0.209]
  BALAM (2-14) | -0.079 [-0.111 to -0.046] | -0.085 [-0.120 to -0.050] | -0.107 [-0.140 to -0.074] | -0.115 [-0.145 to -0.084] | -0.097 [-0.129 to -0.064] | -0.078 [-0.111 to -0.045]

6. Secondary Outcome: Number of Participants Reporting Any Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants reporting any AEs is presented.
Time Frame: Up to Day 15
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 17 | 17 | 15 | 15
Participants | 11 | 14 | 13 | 12 | 15 | 11

7. Secondary Outcome: Number of Participants Reporting Grade >=3 AEs by Preferred Term
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Clinical signs and symptoms that constitute AEs were classified by the investigator as mild (Grade 1), moderate (Grade 2), severe (Grade 3), potentially life threatening (Grade 4), death (Grade 5). Number of participants who experienced grade >=3 AEs by preferred term is presented.
Time Frame: Up to Day 15
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants
  Colitis | 0 | 0 | 1 | 0 | 0 | 0
  Orchitis | 0 | 1 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 3
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 1
  Hypoalbuminaemia | 0 | 0 | 1 | 0 | 0 | 0
  Glycosuria | 0 | 0 | 0 | 1 | 0 | 0
  Orthostatic hypertension | 0 | 0 | 0 | 1 | 0 | 0

8. Secondary Outcome: Number of Participants Reporting AEs (Presented by Severity)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Number of participants reporting Reporting AEs is presented by Severity: Mild- Grade 1 (An event that is usually transient in nature and generally does not interfere with normal activities), Moderate-Grade 2 (An AE that is sufficiently discomforting to interfere with normal activities) and Severe- ≥Grade 3 (An AE that is incapacitating and prevents normal activities). The higher the grade, the more severe the symptoms.
Time Frame: Up to Day 15
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants
  Grade 1 | 6 | 11 | 7 | 6 | 3 | 8
  Grade 2 | 5 | 2 | 5 | 4 | 12 | 0
  >=Grade 3 | 0 | 1 | 1 | 2 | 0 | 3

9. Secondary Outcome: Number of Participants Experiencing AEs Related to Study Intervention
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with use of a study intervention, whether or not considered related to study intervention. An AE is considered related to study intervention if there was a reasonable possibility that the study intervention contributed to the AE.
Time Frame: Up to Day 15
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants | 5 | 3 | 7 | 9 | 15 | 7

10. Secondary Outcome: Number of Participants With Any New Eye Symptom in One or Both Eyes
Description: Eye symptoms were assessed by non-leading questions delivered by trained staff based on a standardized script. A participant with multiple eye symptoms within a preferred term was counted once. Number of participants with any new eye symptom in one or both eyes is presented. All the eye symptoms have been included in the adverse events section of this study.
Time Frame: Up to Day 15
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants | 2 | 5 | 6 | 3 | 10 | 1

11. Secondary Outcome: Average Duration of New Eye Symptom in One or Both Eyes
Description: Average duration of eye symptoms in one or both eyes that were observed after screening for an individual participant was computed as the average duration of all symptoms using the number of symptoms as denominator. Average duration of new eye symptoms in one of both eyes was measured in Hours.
Time Frame: Up to Day 15
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Median (Full Range); unit: Hours
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 2 | 4 | 7 | 7 | 9 | 1
Hours | 12.13 [0.3 to 24.0] | 12.00 [0.1 to 936.0] | 1.79 [0.1 to 336.0] | 72.00 [0.0 to 432.0] | 2.00 [0.1 to 984.0] | 936.00 [936.0 to 936.0]

12. Secondary Outcome: Total Number of Days With New Eye Symptoms in One or Both Eyes
Description: Any day that a participant reported an eye symptom in one or both eyes after screening was counted toward the number of days of having eye symptoms in the study for that participant. Total Number of Days with New Eye Symptoms in One or Both Eyes is presented.
Time Frame: Up to Day 15
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Median (Full Range); unit: Days
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 2 | 4 | 7 | 7 | 9 | 1
Days | 0.51 [0.0 to 1.0] | 0.50 [0.0 to 39.0] | 0.13 [0.0 to 39.1] | 3.00 [0.0 to 34.0] | 0.08 [0.0 to 159.2] | 78.00 [78.0 to 78.0]

13. Secondary Outcome: Change From Baseline in Visual Acuity Score
Description: The visual acuity scores were converted to logarithm to the base 10 of the minimum angle of resolution (logMAR) scale for analyzing change from Baseline. LogMar scale was computed as logMAR = -log(visual acuity score in decimal scale). In logMAR scale, lower scores corresponded to better vision, and as acuity became worse, the value of the logMAR increased. Worst logMAR score was defined to be the highest value of logMAR scores measured on left and right eyes at a given time point. The International Classification of Diseases 11 for distance vision impairment used was: Normal: Equal to or better than 20/40; Mild: Worse than 20/40 and equal to or better than 20/70; Moderate: Worse than 20/70 and equal to or better than 20/200; Severe: Worse than 20/200 and equal to or better than 20/400; Blindness: Worse than 20/400. Baseline was defined as the last assessment at screening. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to Day 15
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Scores on a scale | -0.007 (0.0258) | 0.008 (0.0426) | 0.020 (0.0414) | 0.011 (0.0301) | 0.040 (0.0828) | 0.000 (0.0000)

14. Secondary Outcome: Number of Participants With Color Vision Abnormality in One or Both Eyes
Description: Color vision abnormality was defined as the most severe of protan, deutan, or tritan color deficiency in one or both eyes at a given time point. The degree of severity of color vision deficiency was graded as mild, moderate, severe. The severity of color vision abnormality was assigned to the highest degree of severity of the 3 color vision deficits. Number of participants with color vision abnormality in one or both eyes is presented.
Time Frame: Up to Day 15
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants
  Mild | 2 | 0 | 1 | 2 | 3 | 0
  Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in Heart Rate (HR)
Description: HR was measured twice as follows: after 10 minutes supine ("manual, supine") and after 2 (±0.5) minutes standing ("manual, 2-minute standing"). Baseline was measured on Day 1 before the first dose of study medication was administered. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to Day 15
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
Beats per minute
  Supine HR | 0.6 (9.37) | 0.0 (9.43) | -4.3 (11.30) | -2.8 (11.26) | -2.3 (11.30) | -1.8 (14.16)
  Standing HR | 12.9 (22.20) | 2.3 (16.13) | -5.5 (18.27) | 6.1 (15.53) | -7.4 (12.34) | -3.2 (10.73)

16. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured twice as follows: after 10 minutes supine ("manual, supine") and after 2 (±0.5) minutes standing ("manual, 2-minute standing"). Baseline was measured on Day 1 before the first dose of study medication was administered. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to Day 15
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
Millimeters of mercury (mmHg)
  Supine SBP | -3.0 (16.13) | 0.4 (8.79) | 2.1 (9.74) | -4.1 (9.90) | -4.1 (9.52) | 2.5 (11.14)
  Standing SBP | 2.0 (13.41) | 2.7 (13.85) | 0.6 (10.54) | -2.9 (8.08) | 1.7 (8.15) | 15.7 (16.77)
  Supine DBP | 0.3 (10.69) | 0.1 (7.18) | 1.0 (10.65) | -1.8 (10.89) | -3.7 (6.17) | 2.5 (12.59)
  Standing DBP | 4.9 (8.90) | 2.1 (9.40) | 4.5 (10.99) | -0.1 (7.85) | 1.8 (8.89) | 10.4 (16.19)

17. Secondary Outcome: Change From Baseline in HR as Measured by Electrocardiogram (ECG)
Description: 12-lead ECG was recorded after at least 10 minutes of supine rest to measure HR. Baseline was measured on Day 1 before the first dose of study medication was administered. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Day 15
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
Beats per minute | 2.5 (11.17) | -1.1 (8.91) | -5.8 (9.28) | -2.0 (10.20) | -5.8 (11.37) | -6.0 (10.14)

18. Secondary Outcome: Number of Participants With ≥25% Intraday Increase in HR, ≥25% Intraday Decrease in SBP, ≥25% Intraday Decrease in DBP at Any Intraday Time
Description: HR, SBP and DBP were measured twice as follows: after 10 minutes supine ("manual, supine") and after 2 (±0.5) minutes standing ("manual, 2-minute standing"). Number of participants with ≥25% intraday increase in HR, ≥25% intraday decrease in SBP, ≥25% intraday decrease in DBP at any intraday time is presented.
Time Frame: Day 1 and up to Day 15
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants
  ≥25% increase in supine HR at any intraday time: Day 1 | 5 | 4 | 4 | 3 | 5 | 3
  ≥25% increase in supine HR at any intraday time: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  ≥25% increase in supine HR at any intraday time: Day 15 | 0 | 1 | 0 | 0 | 0 | 1
  ≥25% increase in standing HR at any intraday time: Day 1 | 5 | 2 | 4 | 9 | 4 | 0
  ≥25% increase in standing HR at any intraday time: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  ≥25% increase in standing HR at any intraday time: Day 15 | 2 | 1 | 1 | 3 | 0 | 0
  ≥25% decrease in supine SBP at any intraday time: Day 1 | 0 | 0 | 0 | 0 | 0 | 0
  ≥25% decrease in supine SBP at any intraday time: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  ≥25% decrease in supine SBP at any intraday time: Day 15 | 1 | 0 | 0 | 0 | 0 | 0
  ≥25% decrease in standing SBP at any intraday time: Day 1 | 0 | 0 | 0 | 1 | 1 | 1
  ≥25% decrease in standing SBP at any intraday time: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  ≥25% decrease in standing SBP at any intraday time: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  ≥25% decrease in supine DBP at any intraday time: Day 1 | 0 | 0 | 1 | 1 | 1 | 0
  ≥25% decrease in supine DBP at any intraday time: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  ≥25% decrease in supine DBP at any intraday time: Day 15 | 1 | 0 | 1 | 1 | 0 | 1
  ≥25% decrease in standing DBP at any intraday time: Day 1 | 1 | 1 | 0 | 2 | 1 | 2
  ≥25% decrease in standing DBP at any intraday time: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  ≥25% decrease in standing DBP at any intraday time: Day 15 | 0 | 1 | 0 | 0 | 0 | 0

19. Secondary Outcome: Mean Number of Days With ≥25% Increase in HR From Baseline
Description: HR was measured twice as follows: after 10 minutes supine ("manual, supine") and after 2 (±0.5) minutes standing ("manual, 2-minute standing"). Mean number of days with ≥25% increase in HR from Baseline is presented.
Time Frame: Baseline (Day 1) and up to Day 15
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 9 | 9 | 8 | 12 | 8 | 4
Days
  ≥25% increase in supine HR: number analyzed (Participants) | 9 | 8 | 8 | 9 | 7 | 4
  ≥25% increase in supine HR | 2.3 (1.41) | 4.0 (2.88) | 3.0 (2.07) | 1.8 (1.39) | 4.4 (4.47) | 4.8 (5.50)
  ≥25% increase in standing HR: number analyzed (Participants) | 9 | 9 | 7 | 12 | 8 | 2
  ≥25% increase in standing HR | 5.4 (6.48) | 4.3 (4.80) | 6.1 (4.60) | 3.9 (3.26) | 3.9 (2.70) | 1.0 (0.00)

20. Secondary Outcome: Mean Number of Days With ≥25% Decrease in SBP and Decrease in DBP From Baseline
Description: SBP and DBP were measured twice as follows: after 10 minutes supine ("manual, supine") and after 2 (±0.5) minutes standing ("manual, 2-minute standing"). Mean number of days with ≥25% decrease in SBP and decrease in DBP from Baseline is presented.
Time Frame: Baseline (Day 1) and up to Day 15
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 6 | 2 | 4 | 7 | 5 | 4
Days
  ≥25% decrease in supine SBP: number analyzed (Participants) | 1 | 0 | 2 | 0 | 0 | 0
  ≥25% decrease in supine SBP | 1.0 (NA) — NA indicates that Standard Deviation could not be calculated for 1 participant. |  | 1.0 (0.00) |  |  |
  ≥25% decrease in standing SBP: number analyzed (Participants) | 4 | 1 | 1 | 3 | 2 | 2
  ≥25% decrease in standing SBP | 1.3 (0.50) | 1.0 (NA) — NA indicates that Standard Deviation could not be calculated for 1 participant. | 4.0 (NA) — NA indicates that Standard Deviation could not be calculated for 1 participant. | 1.3 (0.58) | 1.5 (0.71) | 1.0 (0.00)
  ≥25% decrease in supine DBP: number analyzed (Participants) | 4 | 2 | 2 | 4 | 3 | 2
  ≥25% decrease in supine DBP | 1.3 (0.50) | 1.0 (0.00) | 8.0 (9.90) | 2.5 (1.73) | 2.3 (1.15) | 2.0 (0.00)
  ≥25% decrease in standing DBP | 1.3 (0.82) | 2.0 (1.41) | 2.0 (0.82) | 1.9 (1.21) | 1.4 (0.55) | 1.3 (0.50)

21. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters
Description: 12-lead ECG was recorded once at each time point after at least 10 minutes of supine rest to assess PR interval, QRS duration, QT interval, QT Corrected for HR Using Fridericia's Method (QTcF) interval and RR interval. Baseline was measured on Day 1 before the first dose of study medication was administered. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and up to Day 15
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds (ms)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
Milliseconds (ms)
  PR interval: Day 15 | -0.8 (9.06) | -0.7 (6.88) | 0.5 (10.06) | 0.5 (8.10) | 4.1 (15.42) | 2.9 (7.42)
  QRS duration: Day 15 | -0.9 (6.97) | -0.2 (4.63) | 0.1 (8.91) | -0.1 (4.04) | -2.9 (5.84) | 0.8 (6.56)
  QT interval: Day 15 | -3.0 (22.56) | 0.7 (17.89) | 13.4 (20.66) | 9.3 (18.45) | 10.6 (18.90) | 14.2 (20.01)
  QTcF interval: Day 15 | 1.2 (14.68) | -0.8 (10.61) | 7.4 (14.62) | 5.7 (7.15) | 3.1 (9.59) | 6.2 (13.24)
  RR interval: Day 15 | -27.5 (94.60) | 8.4 (83.59) | 41.4 (60.99) | 27.1 (86.48) | 46.6 (100.19) | 52.4 (86.55)

22. Secondary Outcome: Change From Baseline in HR
Description: as for outcome 15
Time Frame: Baseline (Day 1) and at Day 4, Day 7, Day 10 and Day 14
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Beats per minute
  Supine HR: Day 4 | -0.8 (7.59) | 4.2 (10.97) | -0.3 (9.36) | 0.6 (9.41) | -0.8 (10.09) | -3.7 (9.93)
  Standing HR: Day 4 | 6.7 (16.59) | 5.3 (13.40) | -1.8 (20.27) | 3.1 (10.28) | 2.7 (14.06) | -1.5 (7.82)
  Supine HR: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Supine HR: Day 7 | 1.1 (7.58) | -1.0 (8.36) | -5.8 (9.89) | -3.9 (12.35) | -3.5 (8.53) | -9.8 (11.36)
  Standing HR: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Standing HR: Day 7 | 8.7 (20.64) | -3.9 (15.46) | -0.4 (17.41) | 1.4 (14.36) | -4.6 (12.18) | -10.1 (11.47)
  Supine HR: Day 10: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 14
  Supine HR: Day 10 | -2.1 (11.35) | 1.3 (4.30) | -6.0 (10.75) | -3.3 (8.19) | -3.2 (10.39) | -8.5 (11.69)
  Standing HR: Day 10: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 14
  Standing HR: Day 10 | 6.8 (28.37) | 1.7 (10.39) | -6.0 (16.43) | -2.8 (14.57) | -2.5 (13.69) | -11.4 (14.88)
  Supine HR: Day 14: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Supine HR: Day 14 | -3.3 (10.49) | -0.9 (8.82) | -6.4 (12.04) | 0.3 (10.26) | -6.7 (9.62) | -7.1 (14.09)
  Standing HR: Day 14: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Standing HR: Day 14 | 3.1 (18.47) | -0.4 (16.52) | -3.2 (16.92) | 2.1 (13.58) | -9.2 (12.80) | -10.2 (15.15)

23. Secondary Outcome: Change From Baseline in SBP and DBP
Description: as for outcome 16
Time Frame: Baseline (Day 1) and at Day 4, Day 7, Day 10 and Day 14
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Millimeters of mercury (mmHg)
  Supine SBP: Day 4 | -1.3 (9.50) | 0.5 (9.31) | 2.3 (11.13) | -4.2 (7.06) | -2.9 (13.89) | -1.3 (6.53)
  Standing SBP: Day 4 | -0.7 (10.21) | 0.7 (9.04) | -0.4 (8.09) | -4.4 (7.71) | 1.7 (12.30) | 4.3 (10.59)
  Supine SBP: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Supine SBP: Day 7 | -1.7 (10.70) | -3.1 (10.78) | 0.7 (9.19) | -2.2 (12.08) | 0.4 (11.42) | 0.1 (4.94)
  Standing SBP: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Standing SBP: Day 7 | 2.6 (8.63) | 2.0 (10.15) | -3.7 (11.20) | -5.8 (5.89) | -0.3 (10.54) | 5.8 (19.79)
  Supine SBP: Day 10: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 14
  Supine SBP: Day 10 | -4.7 (8.17) | -3.1 (10.65) | 0.9 (9.44) | -2.9 (5.66) | -4.5 (10.46) | -0.5 (8.92)
  Standing SBP: Day 10: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 14
  Standing SBP: Day 10 | -2.3 (11.73) | 3.2 (8.07) | 0.3 (11.12) | -2.3 (6.94) | -1.0 (12.82) | 8.5 (15.24)
  Supine SBP: Day 14: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Supine SBP: Day 14 | -0.5 (5.83) | -1.0 (8.15) | 0.6 (11.44) | -5.3 (10.29) | -1.2 (8.65) | 1.2 (8.90)
  Standing SBP: Day 14: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Standing SBP: Day 14 | 1.5 (11.84) | 5.2 (9.84) | -0.6 (13.00) | -5.1 (8.63) | 1.7 (9.95) | 11.8 (14.82)
  Supine DBP: Day 4 | 1.3 (7.03) | -1.1 (6.74) | -3.0 (12.18) | -1.7 (9.53) | -1.5 (7.35) | -0.4 (5.54)
  Standing DBP: Day 4 | 1.7 (9.23) | -1.5 (4.82) | -3.2 (11.55) | -1.8 (7.87) | 0.4 (10.53) | 6.1 (10.34)
  Supine DBP: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Supine DBP: Day 7 | 0.6 (8.11) | -2.0 (8.68) | -0.5 (9.01) | 1.2 (10.10) | -0.5 (6.76) | 1.4 (7.63)
  Standing DBP: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Standing DBP: Day 7 | 5.1 (7.25) | -0.1 (11.48) | -1.7 (10.97) | -1.5 (7.15) | 1.6 (10.36) | 6.5 (16.58)
  Supine DBP: Day 10: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 14
  Supine DBP: Day 10 | -1.5 (5.97) | -2.6 (5.54) | -1.7 (9.68) | -3.0 (7.39) | -2.1 (6.10) | -0.6 (6.58)
  Standing DBP: Day 10: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 14
  Standing DBP: Day 10 | 2.8 (9.56) | -0.8 (5.73) | 1.9 (7.69) | -1.7 (8.76) | -0.4 (10.45) | 9.4 (13.31)
  Supine DBP: Day 14: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Supine DBP: Day 14 | 0.8 (6.17) | 0.1 (7.07) | -3.1 (10.64) | -2.6 (7.23) | -0.7 (5.68) | 2.5 (7.68)
  Standing DBP: Day 14: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Standing DBP: Day 14 | 2.9 (10.08) | 2.9 (6.66) | 0.9 (11.70) | -1.5 (10.11) | 2.0 (10.62) | 11.8 (14.13)

24. Secondary Outcome: Number of Participants With New Eye Symptoms in Any Eye
Description: Eye symptoms were assessed by non-leading questions delivered by trained staff based on a standardized script. A participant with multiple eye symptoms within a preferred term was counted once. Severe eye symptoms were events with grade 3 intensity or greater. Number of participants with new eye symptoms in any eye including: any, severe and serious is presented.
Time Frame: Day 1, Day 4, Day 7, Day 10, Day 14 and 15
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 1 | 4 | 4 | 2 | 8 | 1
Participants
  Any: Day 1: number analyzed (Participants) | 1 | 0 | 4 | 1 | 8 | 0
  Any: Day 1 | 1 | 0 | 4 | 1 | 8 | 0
  Severe: Day 1: number analyzed (Participants) | 1 | 0 | 4 | 1 | 8 | 0
  Severe: Day 1 | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Day 1: number analyzed (Participants) | 1 | 0 | 4 | 1 | 8 | 0
  Serious: Day 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any: Day 4: number analyzed (Participants) | 0 | 4 | 4 | 2 | 2 | 0
  Any: Day 4 | 0 | 4 | 4 | 2 | 2 | 0
  Severe: Day 4: number analyzed (Participants) | 0 | 4 | 4 | 2 | 2 | 0
  Severe: Day 4 | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Day 4: number analyzed (Participants) | 0 | 4 | 4 | 2 | 2 | 0
  Serious: Day 4 | 0 | 0 | 0 | 0 | 0 | 0
  Any: Day 7: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Any: Day 7 | 0 | 0 | 1 | 0 | 1 | 0
  Severe: Day 7: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Severe: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Day 7: number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0
  Serious: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Any: Day 10: number analyzed (Participants) | 1 | 1 | 0 | 0 | 2 | 1
  Any: Day 10 | 1 | 1 | 0 | 0 | 2 | 1
  Severe: Day 10: number analyzed (Participants) | 1 | 1 | 0 | 0 | 2 | 1
  Severe: Day 10 | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Day 10: number analyzed (Participants) | 1 | 1 | 0 | 0 | 2 | 1
  Serious: Day 10 | 0 | 0 | 0 | 0 | 0 | 0
  Any: Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Any: Day 14 | 0 | 0 | 0 | 0 | 1 | 1
  Severe: Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Severe: Day 14 | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Serious: Day 14 | 0 | 0 | 0 | 0 | 0 | 0
  Any: Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Any: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Severe: Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Severe: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Serious: Day 15 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Change From Baseline in Visual Acuity Score
Description: The visual acuity scores were converted to logMAR scale for analyzing change from Baseline. LogMar scale was computed as logMAR = -log(visual acuity score in decimal scale). In logMAR scale, lower scores corresponded to better vision, and as acuity became worse, the value of the logMAR increased. Worst logMAR score was defined to be the highest value of logMAR scores measured on left and right eyes at a given time point. The International Classification of Diseases 11 classification for distance vision impairment used was: Normal: Equal to or better than 20/40; Mild: Worse than 20/40 and equal to or better than 20/70; Moderate: Worse than 20/70 and equal to or better than 20/200; Severe: Worse than 20/200 and equal to or better than 20/400; Blindness: Worse than 20/400. Baseline was defined as the last assessment at screening. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline, Day 1, Day 4, Day 7, Day 10 and Day 14
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Scores on a scale
  Day 1 | -0.007 (0.0258) | -0.005 (0.0431) | 0.000 (0.0378) | -0.006 (0.0243) | 0.013 (0.0352) | 0.000 (0.0000)
  Day 4 | -0.007 (0.0258) | -0.012 (0.0319) | -0.013 (0.0352) | 0.011 (0.0301) | 0.000 (0.0000) | -0.007 (0.0258)
  Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Day 7 | -0.013 (0.0352) | -0.007 (0.0267) | -0.013 (0.0352) | 0.005 (0.0194) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 10: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 14
  Day 10 | -0.013 (0.0352) | 0.007 (0.0267) | -0.007 (0.0475) | -0.008 (0.0426) | 0.000 (0.0000) | 0.000 (0.0000)
  Day 14: number analyzed (Participants) | 14 | 14 | 14 | 15 | 15 | 13
  Day 14 | -0.014 (0.0363) | 0.000 (0.0392) | 0.007 (0.0475) | -0.013 (0.0352) | 0.000 (0.0000) | 0.000 (0.0000)

26. Secondary Outcome: Number of Participants With Color Vision Abnormality in One or Both Eyes
Description: as for outcome 14
Time Frame: Day 1, Day 4, Day 7, Day 10 and Day 14
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants
  Day 1: Mild: number analyzed (Participants) | 14 | 15 | 15 | 17 | 15 | 15
  Day 1: Mild | 0 | 0 | 1 | 2 | 1 | 0
  Day 1: Moderate: number analyzed (Participants) | 14 | 15 | 15 | 17 | 15 | 15
  Day 1: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Day 1: Severe: number analyzed (Participants) | 14 | 15 | 15 | 17 | 15 | 15
  Day 1: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Day 4: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 7: Mild: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Day 7: Mild | 1 | 0 | 0 | 0 | 1 | 0
  Day 7: Moderate: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Day 7: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Day 7: Severe: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Day 7: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: Mild: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 14
  Day 10: Mild | 0 | 0 | 0 | 0 | 1 | 0
  Day 10: Moderate: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 14
  Day 10: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Day 10: Severe: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 14
  Day 10: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Day 14: Mild: number analyzed (Participants) | 14 | 14 | 14 | 15 | 15 | 13
  Day 14: Mild | 1 | 0 | 0 | 0 | 0 | 0
  Day 14: Moderate: number analyzed (Participants) | 14 | 14 | 14 | 15 | 15 | 13
  Day 14: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Day 14: Severe: number analyzed (Participants) | 14 | 14 | 14 | 15 | 15 | 13
  Day 14: Severe | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Change From Baseline in HR
Description: as for outcome 15
Time Frame: Baseline and at Day 28 and Day 42
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
Beats per minute
  Supine HR: Day 28 | -2.5 (13.10) | -3.6 (17.61) | 0.3 (10.22) | -0.6 (12.90) | 0.8 (15.84) | -4.7 (9.90)
  Standing HR: Day 28: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15 | 14
  Standing HR: Day 28 | 1.3 (23.25) | -9.3 (22.73) | -0.6 (15.22) | 1.2 (15.40) | -3.6 (17.81) | -12.0 (12.65)
  Supine HR: Day 42 | -8.0 (12.12) | 3.9 (12.53) | -3.0 (12.67) | -4.5 (13.57) | -2.3 (17.06) | -9.3 (13.53)
  Standing HR: Day 42: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15 | 14
  Standing HR: Day 42 | -4.4 (22.60) | 0.2 (16.94) | -9.5 (21.00) | -7.1 (9.93) | -11.3 (20.36) | -17.1 (8.59)

28. Secondary Outcome: Change From Baseline in SBP and DBP
Description: as for outcome 16
Time Frame: Baseline and at Day 28 and Day 42
Population: Safety Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
Millimeters of mercury (mmHg)
  Supine SBP: Day 28 | 0.8 (12.52) | 9.2 (11.35) | 7.9 (9.63) | 9.2 (14.22) | -0.1 (11.95) | 6.9 (12.61)
  Standing SBP: Day 28: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15 | 14
  Standing SBP: Day 28 | 3.0 (11.00) | 15.5 (21.20) | 3.7 (13.27) | 10.2 (12.76) | 2.7 (12.98) | 15.7 (17.60)
  Supine SBP: Day 42 | 0.4 (10.51) | 10.0 (10.91) | 2.3 (13.22) | 4.6 (11.71) | 1.9 (11.16) | 6.0 (10.24)
  Standing SBP: Day 42: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15 | 14
  Standing SBP: Day 42 | 3.2 (11.61) | 9.7 (13.17) | 1.1 (11.05) | 9.1 (11.28) | 5.3 (14.14) | 11.9 (17.51)
  Supine DBP: Day 28 | 2.7 (9.66) | 5.2 (8.41) | 5.6 (9.61) | 6.9 (8.94) | 2.5 (6.91) | 6.3 (10.27)
  Standing DBP: Day 28: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15 | 14
  Standing DBP: Day 28 | 8.5 (10.11) | 8.8 (11.15) | 2.7 (10.89) | 9.2 (12.73) | 6.1 (8.93) | 11.8 (15.13)
  Supine DBP: Day 42 | 1.4 (8.02) | 6.1 (6.83) | -1.3 (11.04) | 3.6 (10.78) | 3.3 (7.66) | 2.4 (8.05)
  Standing DBP: Day 42: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15 | 14
  Standing DBP: Day 42 | 8.1 (10.80) | 4.4 (7.54) | -3.5 (8.94) | 7.4 (9.63) | 6.7 (10.51) | 10.1 (12.16)

29. Secondary Outcome: Change From Baseline in Visual Acuity Score
Description: as for outcome 25
Time Frame: Baseline and up to Day 42
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Scores on a scale | -0.007 (0.0258) | 0.000 (0.0302) | -0.007 (0.0458) | -0.006 (0.0429) | 0.000 (0.0000) | 0.000 (0.0000)

30. Secondary Outcome: Number of Participants With Color Vision Abnormality in One or Both Eyes
Description: as for outcome 14
Time Frame: Up to Day 42
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants
  Mild | 0 | 0 | 0 | 0 | 0 | 0
  Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0

31. Secondary Outcome: Number of Participants With Shift From Baseline in Hematology Parameters
Description: Blood samples were collected from participants for analysis of following hematology parameters: Erythrocytes, Hemoglobin, Hematocrit, Leukocytes, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils and Platelets. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, were recorded in the 'To Normal or No Change' category. Baseline was defined as the last assessment at screening. Only the abnormal values were reported where normal to high and normal to low changes were reported.
Time Frame: Day 3, Day 7, Day 15 and Day 42
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants
  Erythrocytes: Normal to Low: Day 3 | 0 | 1 | 0 | 5 | 3 | 2
  Erythrocytes: Normal to High: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Erythrocytes: Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Erythrocytes: Normal to Low: Day 7 | 2 | 1 | 0 | 3 | 3 | 2
  Erythrocytes: Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Erythrocytes: Normal to High: Day 7 | 0 | 0 | 0 | 0 | 0 | 1
  Erythrocytes: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 17 | 14 | 13
  Erythrocytes: Normal to Low: Day 15 | 0 | 1 | 0 | 2 | 3 | 0
  Erythrocytes: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 17 | 14 | 13
  Erythrocytes: Normal to High: Day 15 | 0 | 0 | 0 | 0 | 0 | 1
  Erythrocytes: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Erythrocytes: Normal to Low: Day 42 | 0 | 1 | 0 | 0 | 0 | 2
  Erythrocytes: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Erythrocytes: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 0 | 1
  Hemoglobin: Normal to Low: Day 3 | 3 | 0 | 2 | 3 | 4 | 2
  Hemoglobin: Normal to High: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Hemoglobin: Normal to Low: Day 7 | 3 | 1 | 1 | 2 | 3 | 1
  Hemoglobin: Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Hemoglobin: Normal to High: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Hemoglobin: Normal to Low: Day 15 | 2 | 0 | 1 | 0 | 4 | 0
  Hemoglobin: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Hemoglobin: Normal to High: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Hemoglobin: Normal to Low: Day 42 | 0 | 0 | 0 | 0 | 2 | 1
  Hemoglobin: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Hemoglobin: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit: Normal to Low: Day 3 | 3 | 1 | 2 | 7 | 3 | 1
  Hematocrit: Normal to High: Day 3 | 0 | 0 | 0 | 0 | 0 | 1
  Hematocrit: Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Hematocrit: Normal to Low: Day 7 | 3 | 1 | 2 | 7 | 3 | 0
  Hematocrit: Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Hematocrit: Normal to High: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Hematocrit: Normal to Low: Day 15 | 2 | 0 | 0 | 3 | 3 | 0
  Hematocrit: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Hematocrit: Normal to High: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Hematocrit: Normal to Low: Day 42 | 0 | 0 | 0 | 1 | 2 | 2
  Hematocrit: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Hematocrit: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Normal to Low: Day 3 | 0 | 0 | 1 | 0 | 1 | 1
  Leukocytes: Normal to High: Day 3 | 0 | 1 | 2 | 2 | 4 | 0
  Leukocytes: Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Leukocytes: Normal to Low: Day 7 | 0 | 1 | 0 | 0 | 0 | 0
  Leukocytes: Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Leukocytes: Normal to High: Day 7 | 2 | 0 | 0 | 0 | 0 | 0
  Leukocytes: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Leukocytes: Normal to Low: Day 15 | 1 | 0 | 1 | 0 | 0 | 1
  Leukocytes: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Leukocytes: Normal to High: Day 15 | 0 | 0 | 0 | 0 | 1 | 1
  Leukocytes: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Leukocytes: Normal to Low: Day 42 | 1 | 0 | 0 | 2 | 0 | 2
  Leukocytes: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Leukocytes: Normal to High: Day 42 | 1 | 0 | 1 | 0 | 0 | 0
  Neutrophils: Normal to Low: Day 3 | 1 | 0 | 0 | 0 | 1 | 1
  Neutrophils: Normal to High: Day 3 | 2 | 2 | 1 | 2 | 3 | 0
  Neutrophils: Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Neutrophils: Normal to Low: Day 7 | 0 | 1 | 0 | 0 | 0 | 0
  Neutrophils: Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Neutrophils: Normal to High: Day 7 | 2 | 1 | 1 | 1 | 1 | 1
  Neutrophils: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Neutrophils: Normal to Low: Day 15 | 1 | 0 | 0 | 0 | 0 | 1
  Neutrophils: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Neutrophils: Normal to High: Day 15 | 1 | 1 | 1 | 3 | 0 | 1
  Neutrophils: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Neutrophils: Normal to Low: Day 42 | 1 | 0 | 0 | 0 | 0 | 2
  Neutrophils: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Neutrophils: Normal to High: Day 42 | 0 | 1 | 0 | 0 | 0 | 0
  Lymphocytes: Normal to Low: Day 3 | 0 | 1 | 1 | 1 | 1 | 0
  Lymphocytes: Normal to High: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Lymphocytes: Normal to Low: Day 7 | 0 | 0 | 0 | 1 | 1 | 0
  Lymphocytes: Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Lymphocytes: Normal to High: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Lymphocytes: Normal to Low: Day 15 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocytes: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Lymphocytes: Normal to High: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Lymphocytes: Normal to Low: Day 42 | 0 | 2 | 1 | 1 | 3 | 1
  Lymphocytes: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Lymphocytes: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Normal to Low: Day 3 | 0 | 0 | 0 | 0 | 0 | 1
  Monocytes: Normal to High: Day 3 | 0 | 3 | 6 | 3 | 5 | 0
  Monocytes: Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Monocytes: Normal to Low: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Monocytes: Normal to High: Day 7 | 2 | 3 | 3 | 0 | 1 | 0
  Monocytes: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Monocytes: Normal to Low: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Monocytes: Normal to High: Day 15 | 1 | 1 | 2 | 0 | 0 | 0
  Monocytes: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Monocytes: Normal to Low: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Monocytes: Normal to High: Day 42 | 0 | 0 | 1 | 0 | 1 | 0
  Eosinophils: Normal to Low: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Normal to High: Day 3 | 2 | 1 | 0 | 0 | 0 | 1
  Eosinophils: Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Eosinophils: Normal to Low: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Eosinophils: Normal to High: Day 7 | 2 | 1 | 0 | 0 | 0 | 3
  Eosinophils: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Eosinophils: Normal to Low: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Eosinophils: Normal to High: Day 15 | 3 | 1 | 0 | 0 | 0 | 0
  Eosinophils: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Eosinophils: Normal to Low: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Eosinophils: Normal to High: Day 42 | 3 | 0 | 0 | 1 | 1 | 0
  Basophils: Normal to Low: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Normal to High: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Basophils: Normal to Low: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Basophils: Normal to High: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Basophils: Normal to Low: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Basophils: Normal to High: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Basophils: Normal to Low: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Basophils: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Normal to Low: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Normal to High: Day 3 | 1 | 1 | 2 | 3 | 2 | 3
  Platelets: Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Platelets: Normal to Low: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 14 | 17 | 15 | 14
  Platelets: Normal to High: Day 7 | 3 | 2 | 1 | 4 | 0 | 2
  Platelets: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Platelets: Normal to Low: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Platelets: Normal to High: Day 15 | 1 | 2 | 1 | 2 | 2 | 0
  Platelets: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Platelets: Normal to Low: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Platelets: Normal to High: Day 42 | 0 | 0 | 1 | 0 | 1 | 0

32. Secondary Outcome: Number of Participants With Shift From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected from participants for analysis of following hematology parameters; Alanine Aminotransferase, Aspartate Aminotransferase, Alkaline Phosphatase, Bilirubin, Creatinine, Urea Nitrogen, Sodium and Potassium. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, were recorded in the 'To Normal or No Change' category. Baseline was defined as the last assessment at screening. Only the abnormal values were reported where normal to high and normal to low changes were reported.
Time Frame: Day 3, Day 7, Day 15 and Day 42
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants
  Alanine Aminotransferase: Normal to Low: Day 3 | 0 | 0 | 0 | 0 | 0 | 1
  Alanine Aminotransferase: Normal to High: Day 3 | 4 | 2 | 3 | 1 | 3 | 3
  Alanine Aminotransferase: Normal to Low: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Alanine Aminotransferase: Normal to Low: Day 7 | 0 | 0 | 0 | 0 | 0 | 1
  Alanine Aminotransferase: Normal to High: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Alanine Aminotransferase: Normal to High: Day 7 | 4 | 2 | 3 | 3 | 3 | 3
  Alanine Aminotransferase: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Alanine Aminotransferase: Normal to Low: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 14 | 13
  Alanine Aminotransferase: Normal to High: Day 15 | 5 | 1 | 1 | 5 | 3 | 5
  Alanine Aminotransferase: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Alanine Aminotransferase: Normal to Low: Day 42 | 3 | 2 | 1 | 1 | 0 | 1
  Alanine Aminotransferase: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Alanine Aminotransferase: Normal to High: Day 42 | 1 | 1 | 3 | 0 | 1 | 1
  Aspartate Aminotransferase: Normal to Low: Day 3 | 1 | 0 | 0 | 0 | 1 | 1
  Aspartate Aminotransferase: Normal to High: Day 3 | 1 | 1 | 1 | 1 | 3 | 1
  Aspartate Aminotransferase: Normal to Low: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Aspartate Aminotransferase: Normal to Low: Day 7 | 0 | 0 | 0 | 0 | 0 | 1
  Aspartate Aminotransferase: Normal to High: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Aspartate Aminotransferase: Normal to High: Day 7 | 2 | 0 | 0 | 0 | 1 | 3
  Aspartate Aminotransferase: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Aspartate Aminotransferase: Normal to Low: Day 15 | 1 | 0 | 1 | 1 | 0 | 2
  Aspartate Aminotransferase: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Aspartate Aminotransferase: Normal to High: Day 15 | 1 | 0 | 1 | 1 | 1 | 2
  Aspartate Aminotransferase: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Aspartate Aminotransferase: Normal to Low: Day 42 | 0 | 0 | 2 | 0 | 0 | 0
  Aspartate Aminotransferase: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Aspartate Aminotransferase: Normal to High: Day 42 | 1 | 1 | 2 | 0 | 1 | 0
  Alkaline Phosphatase: Normal to Low: Day 3 | 0 | 0 | 0 | 0 | 1 | 0
  Alkaline Phosphatase: Normal to High: Day 3 | 1 | 0 | 0 | 2 | 1 | 2
  Alkaline Phosphatase: Normal to Low: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Alkaline Phosphatase: Normal to Low: Day 7 | 0 | 0 | 0 | 0 | 1 | 0
  Alkaline Phosphatase: Normal to High: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Alkaline Phosphatase: Normal to High: Day 7 | 2 | 3 | 1 | 2 | 0 | 3
  Alkaline Phosphatase: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Alkaline Phosphatase: Normal to Low: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Alkaline Phosphatase: Normal to High: Day 15 | 3 | 2 | 1 | 3 | 0 | 3
  Alkaline Phosphatase: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Alkaline Phosphatase: Normal to Low: Day 42 | 1 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Alkaline Phosphatase: Normal to High: Day 42 | 0 | 1 | 1 | 0 | 0 | 2
  Bilirubin: Normal to Low: Day 3 | 0 | 0 | 3 | 1 | 0 | 0
  Bilirubin: Normal to High: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: Normal to Low: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Bilirubin: Normal to Low: Day 7 | 1 | 0 | 1 | 3 | 3 | 0
  Bilirubin: Normal to High: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Bilirubin: Normal to High: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Bilirubin: Normal to Low: Day 15 | 1 | 1 | 0 | 1 | 0 | 0
  Bilirubin: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Bilirubin: Normal to High: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Bilirubin: Normal to Low: Day 42 | 0 | 0 | 0 | 1 | 0 | 1
  Bilirubin: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Bilirubin: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine: Normal to Low: Day 3 | 0 | 0 | 0 | 0 | 0 | 2
  Creatinine: Normal to High: Day 3 | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine: Normal to Low: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Creatinine: Normal to Low: Day 7 | 1 | 0 | 2 | 1 | 2 | 2
  Creatinine: Normal to High: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Creatinine: Normal to High: Day 7 | 0 | 1 | 0 | 0 | 1 | 0
  Creatinine: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Creatinine: Normal to Low: Day 15 | 0 | 0 | 0 | 1 | 1 | 0
  Creatinine: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Creatinine: Normal to High: Day 15 | 0 | 1 | 0 | 0 | 0 | 0
  Creatinine: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Creatinine: Normal to Low: Day 42 | 0 | 2 | 0 | 1 | 3 | 1
  Creatinine: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Creatinine: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Normal to Low: Day 3 | 0 | 0 | 1 | 1 | 0 | 1
  Urea Nitrogen: Normal to High: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Normal to Low: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Urea Nitrogen: Normal to Low: Day 7 | 2 | 0 | 2 | 3 | 0 | 0
  Urea Nitrogen: Normal to High: Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Urea Nitrogen: Normal to High: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Urea Nitrogen: Normal to Low: Day 15 | 1 | 0 | 0 | 0 | 1 | 0
  Urea Nitrogen: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Urea Nitrogen: Normal to High: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Urea Nitrogen: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Urea Nitrogen: Normal to Low: Day 42 | 1 | 0 | 4 | 2 | 3 | 3
  Urea Nitrogen: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Urea Nitrogen: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Normal to Low: Day 3: number analyzed (Participants) | 11 | 11 | 12 | 16 | 15 | 11
  Sodium: Normal to Low: Day 3 | 2 | 3 | 4 | 3 | 4 | 2
  Sodium: Normal to High: Day 3: number analyzed (Participants) | 11 | 11 | 12 | 16 | 15 | 11
  Sodium: Normal to High: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Normal to Low: Day 7: number analyzed (Participants) | 12 | 9 | 9 | 15 | 15 | 9
  Sodium: Normal to Low: Day 7 | 3 | 1 | 3 | 4 | 3 | 1
  Sodium: Normal to High: Day 7: number analyzed (Participants) | 12 | 9 | 9 | 15 | 15 | 9
  Sodium: Normal to High: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Normal to Low: Day 15: number analyzed (Participants) | 7 | 8 | 8 | 13 | 15 | 8
  Sodium: Normal to Low: Day 15 | 1 | 1 | 3 | 3 | 1 | 1
  Sodium: Normal to High: Day 15: number analyzed (Participants) | 7 | 8 | 8 | 13 | 15 | 8
  Sodium: Normal to High: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium: Normal to Low: Day 42: number analyzed (Participants) | 5 | 8 | 9 | 15 | 15 | 9
  Sodium: Normal to Low: Day 42 | 0 | 1 | 0 | 1 | 1 | 2
  Sodium: Normal to High: Day 42: number analyzed (Participants) | 5 | 8 | 9 | 15 | 15 | 9
  Sodium: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Normal to Low: Day 3: number analyzed (Participants) | 11 | 11 | 12 | 16 | 15 | 11
  Potassium: Normal to Low: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Normal to High: Day 3: number analyzed (Participants) | 11 | 11 | 12 | 16 | 15 | 11
  Potassium: Normal to High: Day 3 | 3 | 4 | 2 | 3 | 5 | 2
  Potassium: Normal to Low: Day 7: number analyzed (Participants) | 12 | 9 | 9 | 15 | 15 | 9
  Potassium: Normal to Low: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Normal to High: Day 7: number analyzed (Participants) | 12 | 9 | 9 | 15 | 15 | 9
  Potassium: Normal to High: Day 7 | 2 | 2 | 3 | 2 | 0 | 2
  Potassium: Normal to Low: Day 15: number analyzed (Participants) | 7 | 8 | 8 | 13 | 15 | 8
  Potassium: Normal to Low: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Normal to High: Day 15: number analyzed (Participants) | 7 | 8 | 8 | 13 | 15 | 8
  Potassium: Normal to High: Day 15 | 0 | 2 | 2 | 3 | 2 | 0
  Potassium: Normal to Low: Day 42: number analyzed (Participants) | 5 | 8 | 9 | 15 | 15 | 9
  Potassium: Normal to Low: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium: Normal to High: Day 42: number analyzed (Participants) | 5 | 8 | 9 | 15 | 15 | 9
  Potassium: Normal to High: Day 42 | 0 | 2 | 0 | 2 | 0 | 1

33. Secondary Outcome: Number of Participants With Shift From Baseline in Serum Coagulation Parameters
Description: Blood samples were collected from participants for analysis of following serum coagulation: Prothrombin time, Activated Partial Thromboplastin Time and Prothrombin International Normalized Ratio. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, were recorded in the 'To Normal or No Change' category. Baseline was defined as the last assessment at screening. Only the abnormal values were reported where normal to high and normal to low changes were reported.
Time Frame: Day 3, Day 7, Day 15 and Day 42
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Participants
  Prothrombin time: Normal to Low: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin time: Normal to High: Day 3 | 1 | 3 | 3 | 1 | 0 | 0
  Prothrombin time: Normal to Low: Day 7: number analyzed (Participants) | 15 | 12 | 15 | 17 | 15 | 14
  Prothrombin time: Normal to Low: Day 7 | 0 | 0 | 0 | 0 | 0 | 2
  Prothrombin time: Normal to High: Day 7: number analyzed (Participants) | 15 | 12 | 15 | 17 | 15 | 14
  Prothrombin time: Normal to High: Day 7 | 0 | 1 | 1 | 0 | 0 | 1
  Prothrombin time: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 13 | 15 | 15 | 13
  Prothrombin time: Normal to Low: Day 15 | 0 | 0 | 0 | 0 | 0 | 1
  Prothrombin time: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 13 | 15 | 15 | 13
  Prothrombin time: Normal to High: Day 15 | 0 | 3 | 0 | 1 | 0 | 1
  Prothrombin time: Normal to Low: Day 42: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Prothrombin time: Normal to Low: Day 42 | 0 | 0 | 0 | 0 | 3 | 0
  Prothrombin time: Normal to High: Day 42: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Prothrombin time: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 1 | 0
  Activated Partial Thromboplastin Time : Normal to Low: Day 3 | 2 | 0 | 0 | 1 | 1 | 1
  Activated Partial Thromboplastin Time : Normal to High: Day 3 | 1 | 2 | 2 | 1 | 2 | 1
  Activated Partial Thromboplastin Time : Normal to Low: Day 7: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15 | 14
  Activated Partial Thromboplastin Time : Normal to Low: Day 7 | 2 | 1 | 2 | 3 | 1 | 1
  Activated Partial Thromboplastin Time : Normal to High: Day 7: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15 | 14
  Activated Partial Thromboplastin Time : Normal to High: Day 7 | 1 | 0 | 0 | 0 | 1 | 1
  Activated Partial Thromboplastin Time: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Activated Partial Thromboplastin Time: Normal to Low: Day 15 | 3 | 2 | 3 | 2 | 0 | 2
  Activated Partial Thromboplastin Time: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 14 | 15 | 15 | 13
  Activated Partial Thromboplastin Time: Normal to High: Day 15 | 1 | 3 | 0 | 1 | 2 | 2
  Activated Partial Thromboplastin Time: Normal to Low: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Activated Partial Thromboplastin Time: Normal to Low: Day 42 | 2 | 3 | 2 | 3 | 1 | 0
  Activated Partial Thromboplastin Time: Normal to High: Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Activated Partial Thromboplastin Time: Normal to High: Day 42 | 1 | 0 | 0 | 0 | 5 | 0
  Prothrombin International Normalized Ratio: Normal to Low: Day 3 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin International Normalized Ratio: Normal to High: Day 3 | 0 | 0 | 1 | 0 | 0 | 0
  Prothrombin International Normalized Ratio: Normal to Low: Day 7: number analyzed (Participants) | 15 | 12 | 15 | 17 | 15 | 14
  Prothrombin International Normalized Ratio: Normal to Low: Day 7 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin International Normalized Ratio: Normal to High: Day 7: number analyzed (Participants) | 15 | 12 | 15 | 17 | 15 | 14
  Prothrombin International Normalized Ratio: Normal to High: Day 7 | 1 | 0 | 0 | 0 | 0 | 0
  Prothrombin International Normalized Ratio: Normal to Low: Day 15: number analyzed (Participants) | 15 | 14 | 13 | 15 | 15 | 13
  Prothrombin International Normalized Ratio: Normal to Low: Day 15 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin International Normalized Ratio: Normal to High: Day 15: number analyzed (Participants) | 15 | 14 | 13 | 15 | 15 | 13
  Prothrombin International Normalized Ratio: Normal to High: Day 15 | 2 | 2 | 0 | 0 | 0 | 0
  Prothrombin International Normalized Ratio: Normal to Low: Day 42: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Prothrombin International Normalized Ratio: Normal to Low: Day 42 | 0 | 0 | 0 | 0 | 0 | 0
  Prothrombin International Normalized Ratio: Normal to High: Day 42: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Prothrombin International Normalized Ratio: Normal to High: Day 42 | 0 | 0 | 0 | 0 | 0 | 0

34. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Urine Specific Gravity
Description: Urine samples were collected to measure urine specific gravity. Baseline was defined as the last assessment at screening. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Day 3, Day 7 and Day 42
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Ratio
  Day 3 | -0.004 (0.006) | -0.006 (0.009) | -0.002 (0.008) | -0.003 (0.008) | -0.001 (0.008) | -0.003 (0.009)
  Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Day 7 | -0.003 (0.005) | -0.003 (0.008) | -0.004 (0.008) | -0.002 (0.008) | -0.004 (0.008) | -0.003 (0.008)
  Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Day 42 | -0.001 (0.006) | -0.001 (0.008) | 0.001 (0.006) | 0.002 (0.006) | 0.004 (0.008) | 0.001 (0.010)

35. Secondary Outcome: Change From Baseline in Urinalysis Parameter: Urine Potential of Hydrogen (pH)
Description: Urine samples were collected to measure urine pH. Baseline was defined as the last assessment at screening. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Day 3, Day 7 and Day 42
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Potential of Hydrogen (pH)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
Number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 15
Potential of Hydrogen (pH)
  Day 3 | 0.5 (1.13) | 0.3 (1.18) | 0.7 (1.22) | 0.0 (1.37) | 0.2 (1.66) | 0.3 (0.98)
  Day 7: number analyzed (Participants) | 15 | 14 | 15 | 17 | 15 | 14
  Day 7 | 0.6 (1.06) | 0.3 (1.38) | 0.9 (1.06) | -0.1 (1.48) | 0.4 (1.35) | 0.6 (0.85)
  Day 42: number analyzed (Participants) | 15 | 15 | 15 | 17 | 15 | 14
  Day 42 | 0.3 (0.70) | -0.3 (1.45) | 0.4 (0.74) | -0.9 (1.22) | -0.4 (1.35) | 0.1 (0.95)

36. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) After Administration of TBA7371
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of TBA7371. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Days 1, 7 and 14
Population: Pharmacokinetic (PK) Population: included all participants who received at least one dose of TBA-7371 and had at least one pair of pre- and post-dose blood samples with measurable concentrations. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD
Number analyzed (Participants) | 15 | 14 | 15 | 17 | 15
Nanograms per milliliter (ng/mL)
  Day 1 | 4913.52 (16.2) | 4868.80 (8.5) | 9629.97 (11.8) | 5061.16 (21.9) | 16769.92 (14.5)
  Day 7: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15
  Day 7 | 5198.53 (17.6) | 5457.19 (17.4) | 8523.96 (18.4) | 6461.33 (20.7) | 16877.34 (13.0)
  Day 14: number analyzed (Participants) | 15 | 13 | 14 | 15 | 15
  Day 14 | 5323.33 (16.5) | 5351.36 (17.7) | 8671.52 (12.4) | 6060.03 (18.3) | 15599.81 (15.3)

37. Secondary Outcome: Time at Maximum Plasma Concentration (Tmax) After Administration of TBA7371
Description: as for outcome 36
Time Frame: Days 1, 7 and 14
Population: PK Population. Only those participants with data available at the specified data points were analyzed
Measure: Median (Full Range); unit: Hours
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD
Number analyzed (Participants) | 15 | 14 | 15 | 17 | 15
Hours
  Day 1 | 1.000 [0.500 to 4.017] | 1.000 [0.500 to 2.417] | 1.000 [0.500 to 3.933] | 1.000 [0.500 to 2.500] | 1.000 [0.500 to 2.533]
  Day 7: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15
  Day 7 | 1.000 [0.500 to 1.000] | 0.983 [0.500 to 2.417] | 1.000 [0.500 to 6.000] | 1.000 [0.500 to 6.917] | 1.000 [0.500 to 2.567]
  Day 14: number analyzed (Participants) | 15 | 13 | 14 | 15 | 15
  Day 14 | 1.000 [0.500 to 1.000] | 0.500 [0.500 to 2.983] | 1.000 [0.500 to 3.033] | 1.000 [0.500 to 2.483] | 1.000 [0.500 to 4.000]

38. Secondary Outcome: Last Quantifiable Concentration (Clast) After Administration of TBA7371
Description: as for outcome 36
Time Frame: Days 1, 7 and 14
Population: PK Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD
Number analyzed (Participants) | 15 | 14 | 15 | 17 | 15
Nanograms per milliliter (ng/mL)
  Day 1 | 730.077 (713.708) | 1443.136 (611.087) | 1323.935 (969.233) | 2341.459 (710.626) | 3675.478 (1882.844)
  Day 7: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15
  Day 7 | 545.313 (336.060) | 993.427 (560.480) | 1240.299 (1059.177) | 2445.429 (1248.061) | 2942.279 (1752.800)
  Day 14: number analyzed (Participants) | 15 | 13 | 14 | 15 | 15
  Day 14 | 609.215 (481.420) | 913.244 (599.243) | 1043.355 (562.379) | 2148.453 (850.006) | 2510.091 (1103.997)

39. Secondary Outcome: Time at Last Quantifiable Concentration (Tlast) After Administration of TBA7371
Description: as for outcome 36
Time Frame: Days 1, 7 and 14
Population: PK Population. Only those participants with data available at the specified data points were analyzed
Measure: Median (Full Range); unit: Hours
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD
Number analyzed (Participants) | 15 | 14 | 15 | 17 | 15
Hours
  Day 1 | 23.933 [23.867 to 23.983] | 11.917 [10.467 to 12.083] | 23.900 [23.667 to 23.983] | 6.917 [6.800 to 6.983] | 23.917 [23.883 to 24.033]
  Day 7: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15
  Day 7 | 16.450 [16.367 to 17.517] | 11.917 [11.833 to 11.950] | 16.417 [16.367 to 16.533] | 6.917 [6.833 to 6.967] | 16.500 [16.333 to 16.633]
  Day 14: number analyzed (Participants) | 15 | 13 | 14 | 15 | 15
  Day 14 | 16.417 [16.367 to 17.517] | 11.917 [11.833 to 11.983] | 16.450 [16.350 to 16.533] | 6.917 [6.750 to 6.933] | 16.500 [16.333 to 16.550]

40. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 Extrapolated to Infinity (AUCinf) After Administration of TBA7371
Description: as for outcome 36
Time Frame: Day 1
Population: PK Population. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter (h*ng/mL)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD
Number analyzed (Participants) | 14 | 14 | 15 | 15 | 15
Hours*nanograms per milliliter (h*ng/mL) | 51913.151 (25.5) | 44922.259 (23.4) | 111041.711 (24.9) | 44095.496 (24.2) | 256358.739 (23.3)

41. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Last Quantifiable Concentration (AUClast) After Administration of TBA7371
Description: as for outcome 36
Time Frame: Days 1, 7 and 14
Population: PK Population. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter (h*ng/mL)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD
Number analyzed (Participants) | 15 | 14 | 15 | 17 | 15
Hours*nanograms per milliliter (h*ng/mL)
  Day 1 | 44912.674 (19.9) | 30784.091 (10.9) | 92918.441 (15.7) | 21893.926 (17.5) | 192193.142 (12.8)
  Day 7: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15
  Day 7 | 33754.808 (20.1) | 30283.336 (20.8) | 61079.440 (26.7) | 26404.542 (21.5) | 131687.234 (13.1)
  Day 14: number analyzed (Participants) | 15 | 13 | 14 | 15 | 15
  Day 14 | 34087.526 (19.1) | 28951.529 (21.5) | 62866.262 (12.1) | 24619.446 (15.6) | 123208.287 (13.5)

42. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Tau (AUCtau) After Administration of TBA7371
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of TBA7371. PK parameters were analyzed using standard non-compartmental analysis. Tau represents the dosing interval of 24 hours.
Time Frame: Days 1, 7 and 14
Population: PK Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter (h*ng/mL)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD
Number analyzed (Participants) | 15 | 14 | 15 | 17 | 15
Hours*nanograms per milliliter (h*ng/mL)
  Day 1 | 44938.373 (19.9) | 31068.093 (11.1) | 93060.286 (15.7) | 22051.648 (17.5) | 192442.015 (12.8)
  Day 7: number analyzed (Participants) | 15 | 13 | 15 | 17 | 15
  Day 7 | 35906.584 (21.6) | 30368.520 (20.9) | 65868.027 (29.5) | 26551.127 (21.6) | 145179.826 (15.9)
  Day 14: number analyzed (Participants) | 13 | 13 | 14 | 15 | 15
  Day 14 | 35470.923 (20.2) | 29016.288 (21.5) | 67309.556 (14.0) | 24778.661 (15.7) | 134863.281 (14.8)

43. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) After Administration of TBA7371
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of TBA7371. PK parameters were analyzed using standard non-compartmental analysis. Mean and standard deviation for Cmin could not be calculated due to high proportion of NQ values (>30% of values were imputed)
Time Frame: Days 7 and 14
Population: PK Population. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD
Number analyzed (Participants) | 15 | 13 | 15 | 17 | 15
Nanograms per milliliter (ng/mL)
  Day 7 | NA (NA) — Mean and standard deviation could not be calculated as data was only available until 16.5 hours post-dose on Day 7. Samples were needed at 24 hours post dose to get the Cmin. | 756.809 (50.5) | NA (NA) — Mean and standard deviation could not be calculated as data was only available until 16.5 hours post-dose on Day 7. Samples were needed at 24 hours post dose to get the Cmin. | 1777.999 (45.5) | NA (NA) — Mean and standard deviation could not be calculated as data was only available until 16.5 hours post-dose on Day 7. Samples were needed at 24 hours post dose to get the Cmin.
  Day 14: number analyzed (Participants) | 15 | 13 | 15 | 15 | 15
  Day 14 | NA (NA) — Mean and standard deviation could not be calculated as data was only available until 16.5 hours post-dose on Day 14. Samples were needed at 24 hours post dose to get the Cmin. | 715.138 (55.6) | NA (NA) — Mean and standard deviation could not be calculated as data was only available until 16.5 hours post-dose on Day 14. Samples were needed at 24 hours post dose to get the Cmin. | 1736.179 (28.8) | NA (NA) — Mean and standard deviation could not be calculated as data was only available until 16.5 hours post-dose on Day 14. Samples were needed at 24 hours post dose to get the Cmin.

44. Secondary Outcome: Half-life (T1/2) After Administration of TBA7371
Description: as for outcome 36
Time Frame: Days 1, 7 and 14
Population: PK Population. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD
Number analyzed (Participants) | 15 | 14 | 15 | 16 | 15
Hours
  Day 1: number analyzed (Participants) | 14 | 14 | 15 | 15 | 15
  Day 1 | 6.855 (28.4) | 6.395 (26.5) | 7.607 (38.7) | 6.700 (22.7) | 10.695 (32.3)
  Day 7: number analyzed (Participants) | 15 | 12 | 15 | 16 | 15
  Day 7 | 4.222 (20.6) | 3.963 (19.0) | 4.355 (30.9) | 4.534 (29.0) | 5.167 (31.2)
  Day 14: number analyzed (Participants) | 13 | 13 | 14 | 13 | 15
  Day 14 | 3.921 (17.5) | 3.715 (26.8) | 4.295 (22.7) | 4.090 (22.0) | 5.049 (25.0)

45. Secondary Outcome: Accumulation Ratio After Administration of TBA7371
Description: as for outcome 36
Time Frame: Days 7 and 14
Population: PK Population. Only those participants with data available at the specified data points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD
Number analyzed (Participants) | 15 | 13 | 15 | 17 | 15
Ratio
  Day 7 | 1.058 (11.9) | 1.118 (18.8) | 0.885 (22.2) | 1.277 (20.2) | 1.006 (19.3)
  Day 14: number analyzed (Participants) | 15 | 13 | 14 | 15 | 15
  Day 14 | 1.083 (12.3) | 1.096 (15.9) | 0.898 (13.5) | 1.237 (17.5) | 0.930 (16.0)

ADVERSE EVENTS:
Time Frame: Day 1 through Day 15
Description: Safety population which included all participants randomly assigned to study intervention and who received at least one dose of the study intervention.
Arm/Group | TBA-7371 100 mg QD | TBA-7371 100 mg BID | TBA-7371 200 mg QD | TBA-7371 100 mg TID | TBA-7371 400 mg QD | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/17 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15 | 1/15 | 0/17 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 14/15 | 13/15 | 12/17 | 15/15 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TBA-7371 100 mg QD (N=15) | TBA-7371 100 mg BID (N=15) | TBA-7371 200 mg QD (N=15) | TBA-7371 100 mg TID (N=17) | TBA-7371 400 mg QD (N=15) | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE) (N=15)
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TBA-7371 100 mg QD (N=15) | TBA-7371 100 mg BID (N=15) | TBA-7371 200 mg QD (N=15) | TBA-7371 100 mg TID (N=17) | TBA-7371 400 mg QD (N=15) | Isoniazid [H] / Rifampicin [R] / Pyrazinamide [Z] / Ethambutol [E] (HRZE) (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 7 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 3 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colour blindness (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 5 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 1 | 2 | 5 | 0
Conjunctival irritation (Eye disorders) | 1 | 2 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 2 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Photokeratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 4 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 4 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Infusion site discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 2 | 2 | 1 | 1 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 2 | 2 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 3 | 3 | 8 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 2 | 1 | 2 | 4
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Libido increased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT04176250/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT04176250/SAP_001.pdf